CLINICAL TRIAL: NCT02885675
Title: An Observational Study of the Correlation Between miRNA in Peripheral Blood and Prognosis in Patients With ARDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jianfeng Xie, Zhongda Hospital, Southeast University, China
Other Study IDs: ARDS miRNA
Record Dates: First submitted 2016-08-25; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: ARDS
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- ARDS
  Interventions: Other: blood sampling
- Healthy control
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — sample no more than 3ml

SUMMARY:
To evaluate the correlation between the value of miRNA related to ARDS and vascular endothelial cell and ARDS severity, vascular endothelial cell damaging degree，mortality in patients with ARDS.

DETAILED DESCRIPTION:
After consulting literature, we obtain 14 miRNAs related to ARDS and vascular endothelial cell(ARDS-VEC-miRNAs) and 2 biomarkers of scathing vascular endothelial.The ARDS-VEC-miRNAs include miR-15a-5p,miR-16-5p,miR-21-5p,miR-24-3p,miR-26a-5p,miR-27a-3p,miR-27b-3p,miR-126-3p,miR-150-5p,miR-146a-5p,miR-155-5p,miR-221-3p,miR-223-3p,miR-320a.The biomarkers of scathing vascular endothelial include vascular cell adhesion molecule-1(VCAM-1),von Willebrand factor(vWF).20 healthy controls and 60 patients diagnose as ARDS in ICU were included in this study.we blood every participants within 24 hours after enrollment and obtain the plasma.Then, we detecte ARDS-VEC-miRNAs,VCAM-1,vWF levels in plasma by real-time quantitative PCR,record the severity of the illness and survival status within 28 days of every patients.Finally,we evaluate the correlation between the value of miRNA related to ARDS and vascular endothelial cell and ARDS severity, vascular endothelial cell damaging degree，mortality in patients with ARDS.

ELIGIBILITY:
Inclusion Criteria:(1)Admitted to ICU, ARDS patients(Berlin criteria), (2)Patients diagnosed ARDS within 24 hours, (3)Patients age between 18 years old and 85 years.

Exclusion Criteria:1)Pregnant women, 2)Patients with malignant tumor, 3)Immunosuppression or immunocompromised patients.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 healthy controls and 60 patients diagnose as ARDS in ICU were included in this study.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
mortality | 28-day

CONTACTS AND LOCATIONS:
Locations (1):
- Zhong-Da hospital, Nanjing, Jiangsu, China